CLINICAL TRIAL: NCT01138332
Title: Stat3 Signaling Pathway Aberrancies in Pediatric AML
Brief Title: Biomarkers in Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B10; COG-AAML10B10 (Other: Children's Oncology Group); CDR0000671489 (Other: Clinical Trials.gov); NCI-2011-02226 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Blotting, Western

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: western blotting
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in tissue samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of ligand-independent phosphorylation of Stat3 in a small cohort of samples from pediatric patients with acute myeloid leukemia including, but not limited to, samples known to express mutated c-kit.
* Measure the level of Stat3 phosphorylation in these samples after stimulation of three key cytokine receptors expressed on hematopoietic cells IL-6R, G-CSFR, and c-kit.

OUTLINE: Cryopreserved samples are analyzed for levels of various components of the Stat3 pathway via western blotting.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* One of the following karyotypes:

  * t(8;21) and WT c-kit
  * t(8;21) and mutant c-kit
  * Normal karyotype

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Correlations between levels of pY-Stat3 and levels of upstream cytokine receptors
Association of constitutive and/or increased pY-Stat3 and c-kit genotype

CONTACTS AND LOCATIONS:
Overall Officials: Michele S. Redell, MD, PhD, Principal Investigator — Texas Children's Cancer Center